CLINICAL TRIAL: NCT02296944
Title: Anatomical and Functional Results of Surgery of the Tympanic Membrane Perforation of the Child
Acronym: PERFOPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 1798756
Record Dates: First submitted 2014-10-22; First posted 2014-11-21 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Tympanic Membrane Perforation; Tempanoplasty
Keywords: Childrens; tempanoplasty; tympanic membrane perforation; retrospective; cohort
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children aged under 7 years old when tympanoplatie: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery
  Interventions: Other: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery
- Children aged 7 to 10 years at the tympanoplatie: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery
  Interventions: Other: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery
- Children aged 11 to 14 years at the tympanoplatie: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery
  Interventions: Other: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery
- Children aged over 14 years at the tympanoplatie: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery
  Interventions: Other: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery

INTERVENTIONS:
Other: Collection of anatomical and functional results in the appearance of the tympanic membrane after surgery

SUMMARY:
This study is a retrospective cohort of patients minors during the operation of cartilage tympanoplasty for tympanic membrane perforation

DETAILED DESCRIPTION:
The investigators hypothesis is that the cartilage tympanoplastie lead to a closure of the tympanic membrane in 95% of cases. But the investigators believe that certain risk factors may influence the anatomical and functional results of tympanoplastie of the child and that their inclusion could improve these results.

For example, young age is not clear so far as a potential risk factor in the few studies analyzing this factor independently. A recommendation of the French Society of ENT surgery tympanic membrane perforation of the Child in 2006 recommended a minimum age of 6 years. However, the level of evidence of articles analyzed was small (it was basically a consensus of experts) and the investigators feel it necessary to study this factor by age (<7 years, 7-10 years, 11-14 years ,> 14 years) on a large cohort to determine the real influence of age on the anatomical and functional results as this may lead to changes in practice.

Similarly, whatever the influence of age in the general population, it could be a key criterion in children who have a particular field leading to prolonged tubal dysfunction (vélopalatines slots and craniofacial malformations), leading to raising the age of surgery tympanic closure: the investigators have for example in 1000 tympanoplasties for perforation, expected recruitment numbers in this study, 50 patients with craniofacial malformation or vélopalatine slot.

The purpose of this study is to investigate the factors influencing the anatomic outcome at one year of cartilage tympanoplastie child.

ELIGIBILITY:
Inclusion Criteria:

* Patient minors during the operation of cartilage tympanoplasty for tympanic membrane perforation (tympanoplasty for this first ear)
* Patient operated between early 1998 and late 2012
* Postoperative audiometry and otoscopy available between 9 and 18 months after surgery

Exclusion Criteria:

* History of tympanoplasty ipsilateral, tympanic membrane perforation associated with épidermose or cholesteatoma
* The holders of the parent or the patient has reached majority informed the doctor of their refusal to data collection.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric ENT Head and Neck Surgery, Necker hospital.
Sampling Method: Non-Probability Sample
Enrollment: 980 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
anatomical result of the appearance of the tympanoplasty (tympanic membrane perforation after surgery) | 12 months (range 9 to 18 months)
  * Closed eardrum
  * Abnormal eardrum perforation residual, ear effusion, progressive retraction cholesteatoma

SECONDARY OUTCOMES:
Factors influencing the functional outcome of the tympanoplasty | 12 months (range 9 to 18 months)
  * mean bone conduction (BC)
  * air conduction (AC)
  * residual air-bone gap (RR = AC-BC). AC, BC and RR means are calculated on an average of four frequencies 0.5, 1, 2, 4 kHz Good functional outcome will be determined by an average RR ≤20 dB. A labyrinthisation be defined by a mean post-op compounded BC over 10 dB or moypostop BC - BC moypréop> 10 dB.
Factors influencing the functional outcome of the tympanoplasty | 36 months ( range 30 to 42 months)
  * mean bone conduction (BC)
  * air conduction (AC)
  * residual air-bone gap (RR = AC-BC). AC, BC and RR means are calculated on an average of four frequencies 0.5, 1, 2, 4 kHz Good functional outcome will be determined by an average RR ≤20 dB. A labyrinthisation be defined by a mean post-op compounded BC over 10 dB or moypostop BC - BC moypréop> 10 dB.
Change anatomical result of the tympanoplasty | 36 months ( range 30 to 42 months)
factors affecting the anatomical and functional results of the tympanoplasty. | 36 months ( range 30 to 42 months)
  * clinical examination by pediatric ENT
  * hearing test

CONTACTS AND LOCATIONS:
Overall Officials: Françoise DENOYELLE, MD, PhD, Principal Investigator — Hospital Necker - Enfants Malades
Locations (1):
- Hospital Necker - Enfants Malades, Paris, France

REFERENCES:
- [Result] Simon F, Thierry B, Rabeony T, Verrier F, Elie C, Loundon N, Leboulanger N, Couloigner V, Garabedian EN, Denoyelle F. Long-term outcomes of cartilage tympanoplasty in 139 ears in children. Clin Otolaryngol. 2021 Nov;46(6):1395-1399. doi: 10.1111/coa.13801. Epub 2021 May 31. No abstract available. PMID 33993647